CLINICAL TRIAL: NCT02368197
Title: Prospective Randomized Trial Comparing Drug Eluting Balloon Versus Conventional Balloon Angioplasty for Recurrent Cephalic Arch Stenosis in Dialysis Fistulas.
Brief Title: Drug Eluting Balloon Angioplasty for Recurrent Cephalic Arch Stenosis in Dialysis Fistulas
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Verstandig, Dr, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEB.cr.il
Record Dates: First submitted 2014-12-09; First posted 2015-02-20 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Dialysis Access Dysfunction
Keywords: dialysis fistula; cephalic arch stenosis; balloon angioplasty; drug eluting balloon
MeSH Terms: interventions — Paclitaxel; Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard balloon angioplasty (Active Comparator): Dilatation of stenosis with standard non drug eluting balloon catheter
  Interventions: Device: Balloon angioplasty (Bard Dorado)
- Drug eluting balloon angioplasty (Experimental): Dilatation of stenosis with paclitaxel eluting balloon catheter
  Interventions: Drug: paclitaxel (Cardionovum Legflow drug eluting balloon)

INTERVENTIONS:
Drug: paclitaxel (Cardionovum Legflow drug eluting balloon) — Elution of paclitaxel from inflated balloon catheter into vessel wall
  Other Names: Cardionovum Legflow drug eluting balloon
  Arms: Drug eluting balloon angioplasty
Device: Balloon angioplasty (Bard Dorado) — Dilatation of cephalic arch venous stenosis by radial force applied by a balloon catheter
  Other Names: Bard Dorado balloon catheter
  Arms: Standard balloon angioplasty

SUMMARY:
This study is designed to compare the safety and efficacy of paclitaxel-eluting balloon (DEB) versus conventional percutaneous transluminal angioplasty (PTA) for the treatment of hemodynamically significant recurrent cephalic arch stenosis in brachial cephalic fistulas in hemodialysis patients.

DETAILED DESCRIPTION:
The cephalic vein constitutes the major outflow conduit for radial- cephalic autogenous accesses and is the sole outflow conduit for brachial- cephalic autogenous accesses. The portion of the cephalic vein that becomes perpendicular in the region of the deltopectoral groove before its confluence with the axillary or subclavian vein,the cephalic arch, is prone to the development of hemodynamically significant stenosis which is usually treated with balloon angioplasty. Unfortunately restenosis due to angioplasty induced intimal hyperplasia is common and periodic repeated angioplasty is necessary to maintain patency.

Paclitaxel is a mitotic inhibitor used in cancer chemotherapy which is used as an antiproliferative agent for the prevention of restenosis (recurrent narrowing) of blood vessels after balloon angioplasty caused by excessive intimal proliferation. It is locally delivered to the wall of the blood vessel during the dilatation using a paclitaxel eluting balloon.

Initial trials with these balloons have shown promising results in peripheral arteries and early encouraging results in dialysis access.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb dialysis access fistula
* Angiographically demonstrated cephalic arch stenosis >50% within 6 months of last angioplasty using a non drug eluting balloon
* Clinical evidence of hemodynamically significant stenosis: strong pulse and weak thrill on physical exam, prolonged bleeding from puncture sites, raised Kt/V, raised dialysis venous pressure

Exclusion Criteria:

* Contrast allergy
* Unable to give informed consent
* Cephalic arch stent or stent graft
* Life expectancy less then 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Restenosis rate | 6 months
  Incidence of >50% stenosis at the treatment site

SECONDARY OUTCOMES:
Post intervention lesion patency | Up to 12 months
  Interval between intervention and the time of the first subsequent intervention at the treatment site

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Background] Liistro F, Grotti S, Porto I, Angioli P, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for the superficial femoral artery: the DEBATE-SFA randomized trial (drug eluting balloon in peripheral intervention for the superficial femoral artery). JACC Cardiovasc Interv. 2013 Dec;6(12):1295-302. doi: 10.1016/j.jcin.2013.07.010. Epub 2013 Nov 13. PMID 24239203
- [Background] Burzotta F, Brancati MF, Trani C, Porto I, Tommasino A, De Maria G, Niccoli G, Leone AM, Coluccia V, Schiavoni G, Crea F. INtimal hyPerplasia evAluated by oCT in de novo COROnary lesions treated by drug-eluting balloon and bare-metal stent (IN-PACT CORO): study protocol for a randomized controlled trial. Trials. 2012 May 6;13:55. doi: 10.1186/1745-6215-13-55. PMID 22559260